CLINICAL TRIAL: NCT05843266
Title: A Study on the Application of the Early Childhood Attention Battery in a Population of Preterms Children
Brief Title: Early Childhood Attention Battery in Preterm Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Ricci Daniela, Principal Investigator Pediatric Neurologist, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4685
Record Dates: First submitted 2023-03-17; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Attention-deficit; Prematurity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aims of this project are:

1. To explore, using the ECAB, if and in which measure the attentional abilities of young preterm children are different from term peers, whom reference data are already published27.
2. To correlate the ECAB results with the "Conner's Teacher, Rating Scale- Revised e Conner's Parent Rating Scale", one of the available diagnostic interview that helps to identify signs of Attention Deficit Hyperactivity Disorder (ADHD) in young children, at the age of 6 years and over.
3. To study individual trajectories of attention pattern and development during age.

ELIGIBILITY:
Inclusion Criteria:

* gestational age (GA) <34 weeks, intellectual functioning with Intelligence Quotient (IQ>70 verified with Wechsler scales performed within 6 months from the ECAB, age at ECAB assessment between 3 years and 5 years 11 months.

Exclusion Criteria:

* presence of major brain lesions, major motor or behavioral disorders, WPPSI-III subtest receptive vocabulary with a scaled score <8.

Ages: 42 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Low risk preterm children
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-06-25 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
attentional abilities of young preterm children | 3 years
  The Early Childhood Attention Battery (ECAB) consists of 8 subtest assessing 3 aspects of attention: selective attention, sustained attention, attentional control. Counting the number of correct answer we get a raw scores (with a different range for each task) that can be translated in a pondered score and in a percentile based on normative data collected on term born children and previously published

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli, Rome, Italy